CLINICAL TRIAL: NCT02886507
Title: Effects of NSK-SD (Nattokinase) on Blood Pressure. A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Effects of NSK-SD (Nattokinase) on Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Collaborators: JBSL-USA Incorporated (Industry)
Responsible Party: Principal Investigator, Gitte Jensen, Ph.D., Research director, Natural Immune Systems Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIS 087-001
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — nattokinase

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSK-SD (nattokinase) (Active Comparator): One capsule (100 mg) nattokinase/day for the 8-week study duration.
  Interventions: Dietary Supplement: NSK-SD (nattokinase)
- Placebo (Placebo Comparator): One capsule placebo/day for the 8-week study duration.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NSK-SD (nattokinase) — Nattokinase is a fibrinolytic enzyme from the fermented soy product natto. Encapsulated 100mg/capsule, excipient include microcrystalline cellulose.
  Arms: NSK-SD (nattokinase)
Dietary Supplement: Placebo — The placebo capsules contain microcrystalline cellulose.
  Arms: Placebo

SUMMARY:
This is a randomized double-blinded placebo-controlled study to evaluate the effects of NSK-SD consumption in subjects with Stage I hypertension.

The study population will be randomized into two groups, where both groups will receive dietary and lifestyle recommendations to help reduce hypertension. One group will receive placebo and the other group NSK-SD for 8 weeks.

The endpoint will be the change in systolic and diastolic blood pressure after 8 weeks of treatment in the two subject groups.

DETAILED DESCRIPTION:
Previous randomized double blinded placebo-controlled studies on the consumption of the fibrinolytic enzyme Nattokinase and NSK-SD is transported across the gut, and has shown multiple effects on vascular health, including fibrinolytic effects and regulation of blood pressure.

A previous study on effects on blood pressure was conducted in an Asian population involving 86 people, where 73 people completed the study requirements (39 in the NSK-SD group, 34 in the placebo group). The data showed statistically significant reduction in both systolic and diastolic blood pressure after consumption of Nattokinase, whereas the changes after consuming placebo were not significantly different from baseline.

The objective of this study is to evaluate the effects of consumption of nattokinase on hypertension in a North American hypertensive population with associated genetic, dietary, and lifestyle factors. This is in extension of, and contrast to, previous studies in Asian populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of both genders;
* Age 18-85 years;
* Elevated blood pressure as identified by:

  * Systolic blood pressure 130mmHg or higher, or diastolic blood pressure 90mmHg or higher;
  * Confirmed on three separate occasions.

Exclusion Criteria:

* Use of Nattokinase-containing supplements within 60 days prior to enrollment;
* Currently on blood pressure medication;
* History of cancer chemotherapy within the last 12 months;
* Significant active uncontrolled disease (such as lymphoma, cirrhosis, nephritis, uncompensated heart failure);
* Consumption of more than an average of 2 standard alcoholic drinks/day (14 drinks per week)
* Currently experiencing intense stressful events/ life changes that would negatively affect compliance;
* Pregnant, nursing, or trying to become pregnant;
* Women not using effective contraception;
* Food allergies related to ingredients in test product.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Reduction of hypertension | Eight weeks

SECONDARY OUTCOMES:
von Willebrand factor | Eight weeks
Plasma renin activity | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gitte S Jensen, PhD, Principal Investigator — NIS Labs

IPD SHARING:
Plan to Share IPD: Yes
Manuscript publication.